CLINICAL TRIAL: NCT04197778
Title: Food Effect Study of DDO-3055 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DDO-3055-102
Record Dates: First submitted 2019-12-03; First posted 2019-12-13 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Anemia in Chronic Kidney Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental)
  Interventions: Drug: DDO-3055 tablet
- group B (Experimental)
  Interventions: Drug: DDO-3055 tablet

INTERVENTIONS:
Drug: DDO-3055 tablet — DDO-3055 tablet, 2 single doses separated by 6 days.

SUMMARY:
The study is a randomized , open-label, two-stage crossover food effect study of single doses of DDO-3055 tablets in healthy subjects. 14 healthy subjects were randomly divided into groups A and B, 7 subjects in each group. Two stage washout period is 6 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male volunteers, aged 18~45.
* 2. Body weight ≥ 50 kg, body mass index (BMI) between 18 to 28.
* 3. Hemoglobin is in the normal range.
* 4. Signed informed consent.

Exclusion Criteria:

* 1. Vital signs, physical examination, laboratory results are abnormal and clinically significant.
* 2. Currently suffering from cardiovascular, liver, kidney, digestive, nervous, blood, thyroid or mental diseases.
* 3. Suspected allergy to the active ingredient or excipient of the experimental drug.
* 4. Have used erythropoietin within 1 month prior to screening or are currently using erythropoietin.
* 5. Had donated blood or blood transfusion within 3 months prior to screening.
* 6. Vein blood collection is difficult or physical condition can not afford blood collection.
* 7. Hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCVAb), Syphilis antibody, human immunodeficiency virus antibody (HIVAb)were positive.
* 8. Average daily smoking ≥5 cigarettes within 3 months before screening; average daily intake of alcohol within one week is more than 15g (15g alcohol is equivalent to 450mL beer or 150mL wine or 50mL low-alcohol liquor);or 2 days before taking the study drug and during the trial take the tobacco and alcohol and caffeinated foods or drinks, and have special dietary requirements and cannot follow a uniform diet.
* 9. 3 months prior to screening involved in any drug or medical device clinical trials, or within 5 half-life of drugs before screening.
* 10. Any health care products, Over-the-counter drugs or prescription drugs that affects the absorption, distribution, metabolism and excretion of the experimental drug was used within 1 month before the administration.
* 11. With a history of drug abuse or screening visit/baseline visit urine drug abuse screening positive.
* 12. Subjects who are unwilling to take contraceptives or who are likely to donate sperm during the trial and within 30 days after administration; or who do not agree to physical contraception during the trial.
* 13. Other conditions in which the study physician considered the subject not suitable for the trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of DDO-3055 | up to 2 days
Maximum plasma concentration (Cmax) of DDO-3055 | up to 2 days
Time to maximum observed serum concentration (Tmax) of DDO-3055 | up to 2 days
Terminal elimination half-life (T1/2) of DDO-3055 | up to 2 days
Apparent total clearance of the drug from plasma after oral administration (CL/F) of DDO-3055 | up to 2 days
Apparent volume of distribution after oral administration (V/F) of DDO-3055 | up to 2 days

SECONDARY OUTCOMES:
Change of endogenous erythropoietin from baseline | up to 2 days
Safety and tolerability | up to 9 days
  Use the incidence and severity of adverse events to assess safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided